CLINICAL TRIAL: NCT00344110
Title: A Randomized, Double-blind, Placebo and Active-controlled, Multicenter, Parallel-group Study Comparing SPP100 (Aliskiren) 150mg to Placebo and to Losartan 50mg to Evaluate Efficacy, Safety and Pharmacokinetics in Patients With Mild to Moderate Essential Hypertension
Brief Title: Study Comparing SPP100 (Aliskiren) 150mg to Placebo and to Losartan 50mg in Patients With Mild to Moderate Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A1301
Record Dates: First submitted 2006-06-22; First posted 2006-06-26 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Hypertension
Keywords: Hypertension, aliskiren, blood pressure, renin
MeSH Terms: conditions — Hypertension | interventions — aliskiren

INTERVENTIONS:
Drug: Aliskiren

SUMMARY:
Assessing efficacy, safety and pharmacokinetics in patients with mild to moderate essential hypertension

ELIGIBILITY:
Inclusion Criteria:

* Age: 20 - 75 years old
* Gender: Male or female
* Status: Outpatients
* Mild to moderate essential hypertension

Exclusion Criteria:

* Pregnant women, lactating mothers, women suspected of being pregnant, or women who wish to be pregnant
* Patients with msSBP >==180 mmHg and/or msDBP >=110 mmHg at Visit 1, 2 or 3
* Patients with or suspected of having secondary hypertension (due to aortic coarctation, primary aldosteronism, etc.)
* Patients suspected of having malignant hypertension

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 20 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 768 (Actual)
Dates: Start 2006-06; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Mean sitting diastolic blood pressure (msDBP) lowering from baseline to the study end to placebo and losartan

SECONDARY OUTCOMES:
Mean sitting systolic pressure (msSBP) lowering from baseline to the study end to placebo and losartan
Successful response; msDBP <90mmHg and/or a reduction of msDBP ≥ 10mmHg
Control rate; msDBP <90mmHg and msSBP<140mmHg
The pharmacokinetics / pharmacodynamics
Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Japan, Study Chair — Novartis Pharmaceuticals, Japan
Locations (1):
- Novartis Pharmaceuticals, Japan, Japan